CLINICAL TRIAL: NCT06421376
Title: Efficacy and Safety of Inductive Chemoimmunotherapy Followed by Chemoradiotherapy With or Without Surgery in Locally Advanced Esophageal Squamous Cell Cancer: a Single-arm, Prospective, Phase II Trial
Brief Title: Induction Chemoimmunotherapy Combined With Chemoradiotherapy in Esophageal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jianjun Qin, Principal Investigator, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC4475
Record Dates: First submitted 2024-05-10; First posted 2024-05-20 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Esophageal Cancer; Immunotherapy; Induction Therapy; Chemoradiotherapy; Surgery
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inductive chemoimmunotherapy+chemoradiotherapy±surgery (Experimental): In this group, the patients were given 2 cycles of inductive therapy of cardonilizumab combined with chemotherapy, followed by concurrent chemoradiotherapy with two cycles of nab-paclitaxel and cisplatin plus radiotherapy of 50-50.4 Gy. After clinical evaluation, surgery was feasible for a part of patients.
  Interventions: Drug: Cardonilizumab; Radiation: Chemoradiotherapy ±immunotherapy; Procedure: Radical surgery

INTERVENTIONS:
Drug: Cardonilizumab — Two cycles of Inductive therapy： nab-paclitaxel 250mg/ m2+cisplatin 75mg/ m2+Cardonilizumab 10mg/kg，ivgtt，3 weeks per cycle for 2 cycles
Radiation: Chemoradiotherapy ±immunotherapy — Chemoradiotherapy ± immunotherapy：
  * PTV: 50-50.4Gy/1.8-2Gy/25-28fractions ②nab-paclitaxel 100mg+cisplatin 25mg/ m2, d1, every 7 days for 3-5 weeks ③Cardonilizumab 10mg/kg，ivgtt，3 weeks per cycle for 2 cycles
Procedure: Radical surgery — Surgery was evaluated after concurrent chemoradiotherapy according to patients willing and the surgeons' assessment. If patients were accessed with unresectable disease after radiotherapy or refused to receive surgery, Cardonilizumab would be administered for 2 years or until disease progression.

SUMMARY:
Although unprecedented advances have been made in the field of esophageal cancer in recent decades, the prognosis for patients with locally advanced esophageal squamous cell carcinoma (ESCC) remains extremely poor, accounting for 30-40% of overall survival at 5 year. In recent years, multimodal treatments have proven to be an appropriate therapeutic approach for locally advanced ESCC. Recently, immunotherapy developed rapidly. The purpose of this study was to observe the efficacy and safety of cardonilizumab combined with chemoradiotherapy in the treatment of locally advanced ESCC.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old；
* Eligible patients were histologically confirmed esophageal squamous cell carcinoma;
* Eligible patients were proven locally advanced ESCC (cT1-2N1-3M0-1, cT3/T4N0-3M0-1, M1 was limited to supraclavicular lymph node metastasis）diagnosed by computed tomography [CT] and/or endoscopic ultrasonography [EUS] according to the American Joint Committee on Cancer (AJCC) 8th edition staging system；
* ECOG PS score: 0~1；
* Main organs and bone marrow function are normal: routine blood tests: hemoglobin (Hb) ≥100g/L ; absolute neutrophil count (NEUT)≥1.5×109/L; platelets (PLT) ≥100×109/L; white blood cell (WBC)≥3.5×109/L,biochemical examination: alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤1.5×UNL; serum total bilirubin (TBIL) ≤1.5×UNL; serum creatinine ( Cr) 1.0×1.5UNL, and BUN≤1.0×UNL;

Exclusion Criteria:

* Those combined with other primary malignant tumors other than esophageal cancer (except cured basal cell carcinoma of the skin and carcinoma in situ of the cervix);
* patients who had previously received other treatments
* At the time of diagnosis, there were distant and hematogenous metastases beyond the supraclavicular lymph node region, including retroperitoneal multiple lymph node metastasis, bone metastasis, brain metastasis, lung metastasis, liver metastasis, malignant pleural effusion and ascites
* Those who already have esophageal perforation or are at high risk of esophageal perforation
* Patients whose tumors invade close to large blood vessels and are at risk of bleeding in the
* there are active infections, such as active tuberculosis and hepatitis
* There are contraindications to immunotherapy.
* Pregnant or lactating women and women of childbearing age do not take reliable contraceptive measures
* Combined with serious cardiovascular diseases, such as uncontrolled heart failure, coronary heart disease, cardiomyopathy, uncontrolled arrhythmia, uncontrolled hypertension, or a history of myocardial infarction within the past 6 months; and those combined with other uncontrolled acute and chronic diseases such as hypertension and diabetes.
* Violation of inclusion and exclusion criteria, or other reasons that the researcher believes cannot continue the study of drug treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Event-free survival | 1-year
  Time from treatment initiation to locoregional or distant recurrence, or death from any cause.

SECONDARY OUTCOMES:
Overall survival | 1-year
  The 1-year OS rate was defined as the proportion of patients who still alive within one year from treatment initiation.
Adverse events | 1-year
  In terms of adverse events of radiation, chemotherapy and immunotherapy
Locoregional recurrence free survival | 1-year
  The 1-year rate was defined as the proportion of patients who did not have any locoregional recurrence from treatment initiation.
Distant metastasis free survival | 1-year
  The 1-year rate was defined as the proportion of patients who did not have any distant metastasis from treatment initiation.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Wang, Principal Investigator — Department of Radiation Oncology, National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences (CAMS) and Peking Union Medical College (PUMC)
Locations (3):
- China (3):
  - Anyang Cancer Hospital, Anyang, Henan
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - Department of Radiation Oncology, National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences (CAMS) and Peking Union Medical College (PUMC), Beijing

IPD SHARING:
Plan to Share IPD: No